CLINICAL TRIAL: NCT05048277
Title: Single Session Consultation for Parents
Acronym: SSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York University (Other)
Responsible Party: Principal Investigator, Dr. Anil Chacko, Anil Chacko, Ph.D., Associate Professor, New York University, New York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2021-5325
Record Dates: First submitted 2021-08-24; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Parents; Stress
Keywords: Single Session Consultation; SSC; Parents; Parental Stress; Parenting; Stress; Stress Disorders; Children; School-Aged Children; Parental Mental Health
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): The intervention will consist of one 60-minute long session conducted through NYU ZOOM. Each session will be between one parent and one study consultant. The session is goal-oriented and solution-focused. During the SSC, consultants will identify the participant's hope for the session and a specific modifiable goal. From this, the consultant will discuss the "smallest-possible step" participants can take toward overcoming their identified problem and work together in creating an Action Plan, which will present three specific actions the participant can take to accomplishing the session's established goals. Following completion of the two-week follow-up assessment, additional resources personalized to participants will also be provided (i.e., referrals for further services and online resources for parents/children). Ultimately, this intervention is a way to potentially jumpstart progress and facilitate hope and agency.
  Interventions: Behavioral: Single Session Consultation

INTERVENTIONS:
Behavioral: Single Session Consultation — Single-Session Consultation (SSC) is a low-intensity, goal-directed, solution-focused counseling service used for treatment of mental health problems. The intervention consists of a 60-minute session conducted through NYU ZOOM, a HIPAA compliant teleconferencing platform. Sessions will be conducted between a parent and a study consultant. The consultant will 1) identify the participant's specific modifiable goal (and associated "hope"); 2) the "smallest-possible step" taken to overcome their problem; and 3) work collaboratively in creating an Action Plan, drawing on their inner abilities and external resources. This intervention does not act as therapy but instead, to potentially jumpstart progress and facilitate hope and agency. Following completion, participants will receive their Action Plan. Additional personalized resources will be provided following completion of the follow-up assessment, which includes referrals for further services and online resources.

SUMMARY:
Single-Session Consultation (SSC) is a rapidly provided, low-intensity, goal-directed counseling service used for treatment of diverse mental health problems. Research on SSC suggests that, for some clients, a single session of counseling (60 minutes) may help reduce clinical distress.

Despite its benefits, SSC has yet to be evaluated as an alternative for parents (18+) of school-age children (5-12 years old) in the United States with elevated stress levels.

The current research aims to evaluate SSC's feasibility, acceptability, and efficacy as an intervention for this population.

First, perceived acceptability (i.e., parents' participation and successful completion, reschedules, and/or cancellations), usefulness, and client satisfaction will be examined. The investigators will also evaluate whether mechanisms of change (e.g, hope, agency), parental (e.g, stress, mental health), and child (e.g, behavior) outcomes, are improved following the SSC.

The investigators expect SSC to be acceptable, for clients to find SSC to be useful, to be satisfied, and experience an increase in hope and agency after the SSC and hypothesize a reduction in stress levels and improvement in mental health among parents. However, the investigators believe behavior outcomes for the child will remain unchanged.

The investigators will recruit parents via online advertisement on social media. Potential participants will complete a screener through Qualtrics to determine eligibility, which includes location in the United States, age (18+), child's age (5-12 years old), preferred language, child's legal guardianship, technology access, and stress levels. Once eligible, participants will provide consent and make an appointment for their SSC.

The 60-minutes-session will be conducted using HIPAA complaint NYU Zoom with Study Consultants. Parents will complete assessments of parental stress, parental mental health, and child behavior to assess mechanisms (i.e., hope, agency) outcomes and measures of usefulness and satisfaction prior and post the SSC, and another 2-week follow-up questionnaire to monitor progress.

Sessions will be recorded for supervision and treatment fidelity purposes. Upon completion, parents will receive an Action Plan, a written record of the discussion, recommendations, and resources.

ELIGIBILITY:
Inclusion Criteria:

1. Adult parents (18+ years old) who are legal guardians of their school-age children (5 to 12 years old)
2. Must have elevated stress levels based on validated measures obtained through parent self-report
3. Parent must reside in the United States
4. Must be English dominant
5. Can access video-based Zoom conference

Exclusion Criteria:

1. Parent has significant cognitive delays that prohibit involvement in SSC
2. Parent expresses significant personal mental health challenges/child abuse during SSC that warrant immediate discontinuation from SSC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Parenting Stress [Fragile Families Aggravation in Parenting Scale (FFAPS)] from Screener to Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Screener, Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The Fragile Families Aggravation in Parenting Scale is a four-item scale completed by parents to assess parenting stress. Items are rated on a scale from strongly agree to strongly disagree, with greater agreement of items relating to higher levels of stress. The FFAPS has been used in longitudinal studies of parenting and family functioning in the United States and is psychometrically validated for parents of preschool-school-age children. This measure will be used to screen for participant eligibility and as an outcome measure.
Change in Positive and Negative Affect Schedule Short Form (PANAS-SF) from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The PANAS -SF is a 10-item self-report measure that assesses positive affect and negative affect in adults. Scores range from 1 (very slightly or not at all) to 5 (extremely). The items correlate with more specific measures of adult mood and anxiety and is often used in research with community samples to assess mental health functioning. The PANAS-SF is psychometrically-validated (Thomas et al., 2007).
Change in Family Empowerment Scale (family subscale) from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The Family Empowerment Scale (FES) is a parent-report measure to specifically assess empowerment in families with children with emotional/behavioral challenges. The "About Your Family" subscale is a six-item subscale that focuses on parents' confidence in managing their family/child. Scores range from 1 (never) to 5 (very often). Higher total scores indicate a higher level of parent empowerment. The FES has been used in intervention studies with parents/families and has strong psychometric properties.
Change in Readiness for Change Scale from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The Readiness for Change Ruler is a three-item parent-report of parents motivation for change. The ruler is based on the motivational interviewing literature and has been adapted for use for a specific population and research questions. Scores range from 0 (not at all confident/important/ready) to 10 (completely confident/important/ready), with scores above a 5 showing that the person is willing to consider change. The ruler was adapted for use with parents who have stress related to parenting.
Change in Beck Hopelessness Scale from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The Beck Hopelessness Scale is a four-item self-report measure assessing adult hopelessness about the future. Scores range from 1 (absolutely disagree) to 4 (absolutely agree), with higher total scores equating to greater levels of hopelessness. The Beck Hopelessness scale is psychometrically valid.
Change in State Hope Scale from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The State Hope Scale offers a brief, internally consistent, and valid self-report measure of ongoing goal-directed thinking of adults. Scores range from 1 (definitely false) to 8 (definitely true), with higher total scores equating to greater levels of agency.
Change in Behavior and Feelings Questionnaire from Baseline to Within 2 Hours of the Intervention to 2-Week Follow Up | Baseline, Within 2 Hours of Intervention, and 2-Week Follow Up
  The Behavior and Feelings Survey (BFS) is a brief, 12-item rating scale designed to facilitate efficient progress-monitoring during youth psychotherapy. It was developed and evaluated in four samples, among youths ages 7-15 years, with results demonstrating a robust factor structure, internal consistency, test-retest reliability, convergent and discriminant validity, and utility for tracking change during youth psychotherapy (Weisz et al., 2019). The BFS offers caregiver-report forms. Items are rated on a scale from 0 (not a problem) to 4 (a very big problem). Three scale scores can be derived: Internalizing Problems (sum of items 1-6), Externalizing Problems (sum of items 7-12), and Total Problems (sum of items 1-12).
Strengths and Difficulties Questionnaire (SDQ) | Screener
  The Strengths and Difficulties Questionnaire (SDQ) is a short behavioral screening questionnaire for children aged 3 to 16. The questionnaire is used to assess children's mental health and can be completed by children and young people themselves, by their parents, or by their teachers. Scores range between not true to somewhat true to certainly true. For this study, parents will complete the 25 attributes/questions from the SDQ. These 25 items are divided between 5 scales: emotional symptoms (5 items), conduct problems (5 items), hyperactivity/inattention (5 items), peer relationship problems (5 items), prosocial behavior (5 items).

IPD SHARING:
Plan to Share IPD: No